CLINICAL TRIAL: NCT01681069
Title: Double-blind, Randomized, Placebo-controlled, Bicentric Clinical Investigation to Evaluate the Safety and Efficacy of IQP-VV-102 in Reducing Body Weight in Overweight and Obese Subjects
Brief Title: Efficacy and Safety of IQP-VV-102 in Weight Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/009712
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQP-VV-102 (Active Comparator): 2 tablets twice a day
  Interventions: Dietary Supplement: IQP-VV-102
- Placebo (Placebo Comparator): 2 tablets twice a day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-VV-102
  Arms: IQP-VV-102
Other: Placebo
  Arms: Placebo

SUMMARY:
Subjects are randomized to either IQP-VV-102 or a matching placebo. Over 12 weeks, the subjects' body weight, body fat and safety parameters are monitored

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* 25 kg/m2 ≤ BMI ≤ 35 kg/m2
* Written informed consent

Exclusion Criteria:

* Known sensitivity to sources of the active ingredients and excipients
* Pregnancy or nursing
* Inability to comply with study requirements, e.g. due to language difficulties
* Participation in another study during the last 30 days of the screening visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grube, MD, Principal Investigator — Practice for General Medicine
Locations (1):
- Barbara Grube, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Grube B, Bongartz U, Alt F. IQP-VV-102, a Novel Proprietary Composition for Weight Reduction: A Double-Blind Randomized Clinical Trial for Evaluation of Efficacy and Safety. Evid Based Complement Alternat Med. 2015;2015:413075. doi: 10.1155/2015/413075. Epub 2015 May 17. PMID 26074990

RESULTS

PARTICIPANT FLOW:
Groups:
- IQP-VV-102: 2 tablets twice a day
  IQP-VV-102
- Placebo: 2 tablets twice a day
  Placebo
Period: Overall Study
Arm/Group | IQP-VV-102 | Placebo
Started | 60 | 60
Full Analysis Set (FAS) | 57 | 60
Completed | 55 (Valid Case Analysis Set (VAS)) | 53 (Valid Case Analysis Set (VAS))
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: *Only 117 out of 118 subjects included in the intention-to-treat population as one subject was lost to follow-up after visit 3
Groups:
- Total: Total of all reporting groups
Arm/Group | IQP-VV-102 | Placebo | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Continuous [Mean (Standard Deviation); unit: year] | 43.6 (11.6) | 40.5 (11.9) | 42.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 12 | 22 | 34
Body Weight [Mean (Standard Deviation); unit: kg] | 82.0 (10.6) | 84.9 (12.9) | 83.5 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight at End of Study Compared to Baseline
Description: Change in body weight at the end of study compared to baseline
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IQP-VV-102 | Placebo
Number analyzed (Participants) | 57 | 60
kg | 3.29 (2.30) | 0.83 (2.00)

2. Secondary Outcome: Change in Waist Circumference (in cm) at End of Study From Baseline
Description: Difference in waist circumference (in cm) at end of study from baseline
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | IQP-VV-102 | Placebo
Number analyzed (Participants) | 57 | 60
cm | 2.11 (2.09) | 0.81 (2.02)

3. Secondary Outcome: Change in Mean Body Fat at End of Study From Baseline
Description: Measured in kg using calibrated weighing scales
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IQP-VV-102 | Placebo
Number analyzed (Participants) | 57 | 60
kg | 2.14 (3.42) | 0.56 (2.43)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: All adverse effect reported were not deemed associated with the investigational product
Arm/Group | IQP-VV-102 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/60
Other Adverse Events (participants affected / at risk) | 5/57 | 8/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQP-VV-102 (N=57) | Placebo (N=60)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory infections (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Vomitting and diarhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypothyrodism (Endocrine disorders) | 1 | 0
Headache (General disorders) | 0 | 3
Bruised left thigh (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other